CLINICAL TRIAL: NCT04494971
Title: Pilot Validation of an App to Estimate and Manage Portion Size: The PortionSize Smartphone App
Brief Title: The PortionSize Smartphone App Pilot (PS Pilot)
Acronym: PS Pilot
Status: Completed | Type: Observational
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Corby K. Martin, PBRC Professor, Director - Ingestive Behavior Laboratory, Pennington Biomedical Research Center
Other Study IDs: PBRC 2019-013
Record Dates: First submitted 2020-07-28; First posted 2020-07-31 (Actual); Results first posted 2024-10-15 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-10

CONDITIONS: Dietary Habits
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective is to examine the preliminary validity, reliability and perceived participant satisfaction of the PortionSize app.

DETAILED DESCRIPTION:
Overweight and obesity are a burgeoning public health concern, yet only a small minority of smartphone apps that claim to facilitate healthy eating and weight loss incorporate evidence-based principles. Such innovations are important as humans fundamentally cannot accurately estimate portion size. Indeed, portion size estimation errors account for ~50% of the error in self-reported food intake, and data from our laboratory has demonstrated that extensive training results in only modest improvements in portion size estimation accuracy and that portion size estimates remain inaccurate. Our long-term goal is to create simple and accessible interventions that assist individuals with weight control. In particular, we aim to provide easy-to-use phone apps that allow participants to monitor the portion sizes of the foods they consume. These apps guide participants on appropriate portion sizes and provide recommendations of food groups that should be consumed. To that end, we have developed the PortionSize app. We propose to improve the accuracy of portion size measurement, as it is poorly determined by self-report measures. This will occur via the development of the PortionSize smartphone app and this pilot study will test the usability as well as preliminary validity and reliability of the app functionality.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18.5-45 kg/m2 based upon self-reported height and weight
* Have an iPhone and an operable Apple ID, password, and email address and is willing to use these to collect data during the study, acknowledging that data usage, and associated charges, are a result of study participation

Exclusion Criteria:

* For females, pregnancy or breast feeding
* Currently diagnosed with an eating disorder
* Disease that severely affects metabolism, including diabetes, hypercholesterolemia, or dyslipidemia
* Has gained or lost more than 10 lbs in the last 3 months
* PBRC faculty/staff member
* Has suffered serious mental illness that has resulted in serious functional impairment and has substantially interfered with one's life activities within the last 5 years
* Any other medical, psychiatric, or behavioral factors in the judgment of the Principle Investigator that may interfere with study participation or the ability to follow the protocol

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Healthy participants ages 18 to 65 in the Baton Rouge, LA area.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2020-08-31 (Actual); Primary Completion 2020-11-20 (Actual); Study Completion 2020-11-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Apolzan, PhD, Principal Investigator — Pennington Biomedical Research Center; James Dorling, PhD, Principal Investigator — Pennington Biomedical Research Center; Corby Martin, PhD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Diktas HE, Lozano CP, Saha S, Broyles ST, Martin CK, Apolzan JW. Evaluating the Validity of the PortionSize Smartphone Application for Estimating Dietary Intake in Free-Living Conditions: A Pilot Study. J Nutr Educ Behav. 2024 Sep;56(9):643-652. doi: 10.1016/j.jneb.2024.05.226. Epub 2024 Jun 18. PMID 38888538

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Cohort: The validity, reliability, and satisfaction of the PortionSize app under controlled and free-living conditions were quantified.
Period: Overall Study
Arm/Group | Study Cohort
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Study Cohort
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | NA — Ages eligible for study were 18 Years to 65 Years
  Between 18 and 65 years | 15
  >=65 years | NA — Ages eligible for study were 18 Years to 65 Years
Age, Continuous [Mean (Standard Deviation); unit: years] | 28 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Validity of Portion Size at Estimating Energy Intake in Laboratory Conditions
Description: Compared measurements from PortionSize to weighed values in the laboratory, which is the criterion measure.
Time Frame: 1 simulated meal collected on one day
Measure: Mean (Standard Deviation); unit: kcal
Groups:
- Study Cohort: The validity of the PortionSize app under controlled (laboratory) conditions was quantified.
Arm/Group | Study Cohort
Number analyzed (Participants) | 15
kcal
  Mean energy intake estimated with the PortionSize app | 742.9 (328)
  Mean energy intake estimated with the directly weighed food portions | 659.3 (190.7)

2. Primary Outcome: Validity of Portion Size at Estimating Energy Intake in Free-living Conditions
Description: Quantify the validity of the app measurements in free-living conditions compared to digital photography (the criterion measure).
Time Frame: Mean kcal intake over 3 days
Measure: Mean (Standard Deviation); unit: kcal
Groups:
- Study Cohort: The validity of the PortionSize app under free-living conditions was quantified.
Arm/Group | Study Cohort
Number analyzed (Participants) | 14
kcal
  Mean energy intake estimated with the PortionSize app | 1560.6 (446.8)
  Mean energy intake estimated with rater analysis of food photos | 1349.7 (389.2)

ADVERSE EVENTS:
Time Frame: 3 months (during the study period)
Description: This study involved no greater than minimal risk.
Arm/Group | Study Cohort
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-08-24): https://cdn.clinicaltrials.gov/large-docs/71/NCT04494971/Prot_SAP_000.pdf
  • Informed Consent Form (2020-08-24): https://cdn.clinicaltrials.gov/large-docs/71/NCT04494971/ICF_001.pdf